CLINICAL TRIAL: NCT01351402
Title: Investigating the Effects of Massage vs. Rest on Oxytocin, ACTH, and B-endorphins
Brief Title: Effects of Massage Versus Rest on Hormones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claremont Graduate University (Other)
Collaborators: Gruter Institute (Unknown)
Responsible Party: Paul J. Zak, Ph.D., Center for Neuroeconomic Studies, Claremont Graduate University
Allocation: Randomized | Masking: Single | Purpose: Basic Science
Other Study IDs: 00012002
Record Dates: First submitted 2011-05-06; First posted 2011-05-10 (Estimated); Last update posted 2011-05-10 (Estimated); Status verified 2005-08

CONDITIONS: Massage; Rest
Keywords: Massage; Rest
MeSH Terms: interventions — Massage; RE1-silencing transcription factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Massage or Rest — Participants either received 15 minutes of moderate pressure Swedish massage on the upper back, or rested quietly sitting in a chair for 15 minutes.

SUMMARY:
This study will investigate the effects of 15 minutes of massage compared to 15 minutes of quiet rest on physiological variables. Specifically, the investigators will measure the effects on levels of the social hormone oxytocin, and on other physiological variables that interact with oxytocin or that may be influenced by massage (including ACTH, Beta-endorphin, and IL-1alpha). The investigators will also investigate whether, in the case of hormones changes, these influence social decision making.

DETAILED DESCRIPTION:
Interested participants will have the experiment explained both verbally and in writing, and asked to give their informed consent in writing. After consent, the participants will be led to a private room for their first 30ml blood draw by a qualified phlebotomist. Participants will then have a second 30ml blood draw.

ELIGIBILITY:
Inclusion Criteria:

* Anyone English speaking and over the age of 18.

Exclusion Criteria:

* Minors and anyone who has used illicit drugs or alcohol in the last 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2006-06; Primary Completion 2006-08 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Oxytocin | Within 5 minutes following experimental manipulation of either 15 minutes massage or rest.
  Participants receive a blood draw at baseline and immediately following 15 minutes of massage or rest and oxytocin will be measured from this sample.

SECONDARY OUTCOMES:
Adrenocorticotrophic hormone (ACTH) | Within 5 minutes following experimental manipulation of either 15 minutes massage or rest.
  Participants will receive a blood draw at baseline and immediately following 15 minutes of massage or rest, and ACTH will be measured in these blood samples.
Beta-endorphin | Within 5 minutes following experimental manipulation of either 15 minutes massage or rest.
  Participants will receive a blood draw at baseline and immediately following 15 minutes of massage or rest, and B-endorphin will be measured from these samples.
Interleukin-1alpha (IL-1a) | Within 5 minutes following experimental manipulation of either 15 minutes massage or rest.
  Participants will receive a blood draw at baseline and immediately following 15 minutes of massage or rest, and IL-1a will be measured from these samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Cassel, UCLA, Los Angeles, California, United States